CLINICAL TRIAL: NCT00204256
Title: Open Randomized Phase IV Study on Intravenous Iron in Anemic Patients With Chronic Kidney Disease
Brief Title: Intravenous Iron in Patients With Anemia of Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ven-PD-03; Iron-Predialysis-2003
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Kidney Failure, Chronic
Keywords: chronic kidney disease; anemia; intravenous iron; recombinant human erythropoetin
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Anemia | interventions — Ferric Oxide, Saccharated

INTERVENTIONS:
Drug: Iron sucrose

SUMMARY:
The objective of this study is the evaluation of the efficacy and safety of intravenous iron sucrose in anemic patients with chronic kidney disease not on renal replacement therapy.

DETAILED DESCRIPTION:
This is a randomized, open label, phase IV study in anemic predialysis patients (Hb between 8 and 11.5 g/dl) who require iron supplementation. The duration of the study for each patient will be approximately 6 months. Patients will be randomized to one of two treatment arms and admitted to the anemia correction phase (days 1-43). Treatment will be intravenous iron sucrose alone versus iron sucrose plus rhEPO. The main treatment evaluation will at the end of the correction phase: The primary end-point will be the change of hemoglobin during correction phase. Secondary end-points will be the change of ferritin and transferrin saturation from baseline to day 43. Safety assessments will include recording of adverse events, vital signs, physical examinations and clinical laboratory tests. Incidence and severity of adverse events will be compared between the two different treatment arms.

ELIGIBILITY:
Inclusion Criteria:

Chronic kidney disease Anemia (Hb 8 - 11.5 g/dl) Age above 18 years Signed informed consent

Exclusion Criteria:

Rapid progression of kidney disease Need for dialysis Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-03; Study Completion 2005-03

PRIMARY OUTCOMES:
Change in hemoglobin from baseline to day 43

SECONDARY OUTCOMES:
Change in ferritin and transferrin saturation from baseline to day 43; incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Roland M Schaefer, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, Westphalia, Germany